CLINICAL TRIAL: NCT02006810
Title: Development of Endothelial Biomarkers for Use in Cohort Studies. Comparison With Reference Biomarkers.
Brief Title: Development of Endothelial Biomarkers
Acronym: NUTREND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHU-0168; 2013-A00205-40
Record Dates: First submitted 2013-09-24; First posted 2013-12-10 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Metabolic Syndrome
Keywords: Endothelium biomarkers; Atherosclerotic disease; Endothelial function; Nutritional stimuli
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- lipids (Experimental): The study will be randomized (on the order of taking the products: a single dose of lipids or a single dose of flavonoids), single-blinded, cross-over for each population (healthy and metabolic syndrome).
  Interventions: Behavioral: Induction of endothelial function variations
- flavonoids (Other): The study will be randomized (on the order of taking the products: a single dose of lipids or a single dose of flavonoids), single-blinded, cross-over for each population (healthy and metabolic syndrome).
  Interventions: Behavioral: Induction of endothelial function variations

INTERVENTIONS:
Behavioral: Induction of endothelial function variations
  Other Names: Improvement with cocoa polyphenol dose; Induction of dysfunction with lipid dose

SUMMARY:
The main objective is to develop and validate new endothelial function markers discriminating and reproducible by assessing the ability to reveal changes in endothelial function in response to positive and negative nutritional stimuli.

DETAILED DESCRIPTION:
The study will be randomized (on the order of taking the products: a single dose of lipids or a single dose of flavonoids), single-blinded, cross-over for each population (healthy and metabolic syndrome).

ELIGIBILITY:
Inclusion Criteria:

* - 40 to 65 years old
* male
* non-smokers

Specific inclusion criteria for healthy subjects :

* Healthy subjects should not take antihypertensive or statin.
* Healthy subjects should not present metabolic syndrome but one criterion of the metabolic syndrome will be tolerated.

Specific inclusion criteria for subjects with metabolic syndrome :

- subjects with metabolic syndrome must have at least 3 of the 5 criteria associated with the metabolic syndrome.

Exclusion Criteria:

* treatment vasodilator nitric oxide liberating,
* diabetes and coronary artery disease,
* chronic alcoholism,
* severe hepatic impairment,
* end stage renal failure or dialysis,
* neurological tremor,
* cancer, mental illness or other severe disease which can impact informed consent and / or results,
* Refusal to be registered in the National File of Volunteers
* Person in exclusion of the National Volunteer File

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Flow Mediated Dilatation (FMD)compared to hyperemic velocity time integral (VTI) and endothelial microparticles (MPE) | at 150 mn after the product intake
  Changes in endothelial function from baseline at 150 mn after the product intake, evaluated by:
  - Flow Mediated Dilatation (FMD) (reference)
  Compared to:
  * Hyperemic Velocity Time Integral (VTI)
  * Endothelial microparticles (MPE)

SECONDARY OUTCOMES:
Changes in endothelial function evaluated by cell adhesion molecule (CAM) and micro-RNA (miRNA) | at 150 mn after the product intake
  Changes in endothelial function from baseline at 150 mn after the product intake, evaluated by:
  * Cell Adhesion Molecule (CAM)
  * Micro-RNA (miRNA)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BARBER CHAMOUX, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France